CLINICAL TRIAL: NCT02660476
Title: Qatar Universal Diabetes Outcomes (QUDOS) Study
Acronym: QUDOS
Status: Terminated | Type: Observational
Why Stopped: The study has been closed by our IRB due to the PI's departure from the Institution.
Sponsor: Weill Cornell Medical College in Qatar (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: JIRB: 14-0032. MRC: #14461/14
Record Dates: First submitted 2015-05-20; First posted 2016-01-21 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: Diet; Middle East and North Africa country; Health; Complication; Cardiovascular disease; Obesity; Stress; Obstructive Sleep Apnoea (OSA)
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine, saliva and stool samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- QUDOS 1: Aims to recruit 1,700 diabetic patients (including 200 with type 1 diabetes mellitus (independent of healthcare setting)) attending the hospitals and primary care
- QUDOS 2: To further characterise 500 patients, from the total 1500 patients with T2DM recruited in QUDOS 1, who accept to continue with QUDOS 2 (a more detailed study and assessment).

SUMMARY:
QUDOS is a cross-sectional population study aiming to answer key questions about diabetes and its complications in Qatar as well as identify factors associated with the development and progression of diabetes complications.

DETAILED DESCRIPTION:
QUDOS aims to gain a better understanding of diabetes in primary and secondary care over a period of 24 months.

A range of patients with diabetes will be sampled (including those with Type 1 diabetes as this group is under-studied in Qatar). This will be important in designing appropriate intervention plans that will improve diabetic patients' health conditions to prevent or delay the onset of complications and will provide a strong foundation for longitudinal study.

The broad objectives of the study are:

QUDOS 1: Aims to recruit 1,700 diabetic patients (including 200 with type 1 diabetes mellitus (independent of healthcare setting)) attending the hospitals and primary care and to collect the following data:

* Demographics: age, sex, ethnicity, socio-economic background, smoking status;
* Anthropometrics: vital signs, height, weight, body fat percentage, fat mass, neck and waist circumference;
* Medical History: medications, complications, comorbidities, latest HbA1c and lipid profiles and family medical history;
* Routine laboratory data;
* Lifestyle: diet, physical activity,;
* Sleep: quality and daytime sleepiness;
* Cognition and Mental Health: depression, anxiety, stress and memory;
* Diabetes microvascular complications: diabetic neuropathy, urine albumin/creatinine ratio; routine retinal screening data.
* Gut microbiome from a stool sample

QUDOS 2: To further characterise 500 patients, from the total 1500 patients with T2DM recruited in QUDOS 1, who accept to continue with QUDOS 2 (a more detailed study and assessment).

This phase aims to concentrate on the following aspects:

* Obstructive sleep apnoea;
* Sleep duration and quality;
* Diet;
* Objective physical activity;
* Stress;
* Quality of Life;
* Depression and anxiety;
* Perceived control of health;
* Detailed neuropathy screening;
* Cardiovascular function;
* Cognitive function;
* Biological samples.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 and Type 2 diabetes mellitus;
2. Male or Female;
3. Resident in Qatar;
4. MENA birthplace and family origin;
5. 18-70 years old;
6. Capable to give informed consent and complete the study.

Exclusion Criteria:

1. Known pregnancy or planning pregnancy during the duration of study; 2. Congenital disorders; 3. Terminal illness; 4. Enrolled in a clinical trial involving medication; 5. Uncontrolled mental illness preventing participation; 6. Those who have already experienced a definitive microvascular complication:

i. End-stage renal disease; ii. Major amputation; iii. Blindness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18-70 years old with diabetes, who are a resident in Qatar or born in one of the MENA countries with family originating from MENA countries, will be recruited from one of the following sites:
  * Primary health care centers
  * Hamad General Hospital
  * Al-Wakra Hospital
  * Al-Khor Hospital
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2014-10; Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Diabetes Complications (Nephropathy, Neuropathy, Retinopathy) | Baseline (Cross-Sectional)
  Our primary analyses will be conducted to explore the potential cross-sectional relationships amongst proposed factors related to type 2 diabetes complications

SECONDARY OUTCOMES:
Mental Health | Baseline (Cross-Sectional)
  To assess the relationships between T2DM and depression through questionnaires
Sleep and sleep related breathing disorders | Baseline (Cross-Sectional)
  To assess the relationships between T2DM and sleep disordered breathing, sleep duration and sleep quality through a home sleep study
Physical activity | Baseline (Cross-Sectional)
  To assess the relationships between T2DM and physical activity using an Actiwatch

CONTACTS AND LOCATIONS:
Overall Officials: Shahrad Taheri, PhD, Principal Investigator — Weill Cornell Medical College in Qatar
Locations (1):
- Weill Cornell Medicine Qatar, Doha, Qatar